CLINICAL TRIAL: NCT00949234
Title: A Pilot Project to Operationalize the Prevention Strategy of Post Exposure Prophylaxis Following Sexual Exposure to HIV in Combination With Educational Programming and Behavioral Risk Reduction Strategies in Los Angeles County
Brief Title: Interventions for HIV Negative Men and Women Who Have High-risk Suspected Exposure to HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Los Angeles County Department of Public Health (Other Government); AIDS Project Los Angeles (Other); Los Angeles LGBT Center (Other); The OASIS Clinic (Unknown)
Responsible Party: Principal Investigator, Dr. Raphael Landovitz, Associate Director, UCLA Center for Clinical AIDS Research & Education (CARE), University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PQUAD
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: HIV Prevention; HIV Infections
Keywords: post exposure prophylaxis; biomedical prevention; HIV seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; Lopinavir; Ritonavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-Label (Other): This was an open-label demonstration project. Therefore, medications were not blinded and participants were made aware of the regimen they received for PEP.
  Interventions: Drug: tenofovir + emtricitabine, lopinavir/ritonavir

INTERVENTIONS:
Drug: tenofovir + emtricitabine, lopinavir/ritonavir — The preferred regimen will be tenofovir + emtricitabine, provided as a fixed-dose combination tablet as Truvada®. Dosing is 1 tablet by mouth once daily. For participants with a creatinine clearance 30-49 mL/min, dosing of Truvada is 1 tablet by mouth every other day. For patients with creatinine clearance <30 mL/min or on hemodialysis, Truvada should not be used. For intolerance to Truvada, Combivir (zidovudine 300mg/lamivudine 150mg)will be available to be taken as 1 PO BID. For highest-risk category exposures (receptive anal intercourse with a known or suspected HIV-positive source patient or in cases of suspected source drug resistance, see Schema, below) one of the following should be added to the above "standard" treatment, creating an "expanded" regimen:
  Preferred: Lopinavir/ritonavir (200mg/50mg), 2 tablets orally twice daily or 4 tablets once daily
  Other Names: Truvada; Combivir

SUMMARY:
The purpose of this program is to evaluate an effort to provide a comprehensive package of HIV prevention services of which post-exposure prophylaxis (medicines that may help prevent HIV infection after an exposure) can be a part. It will also include risk reduction information and testing for other sexually transmitted infections.

DETAILED DESCRIPTION:
The Los Angeles County P-QUAD program is a combined effort of County, City, public health, community, academic, and private agencies and individuals in an effort to provide a comprehensive package of HIV prevention services of which PEP can be an integral component. These services are designed to be easily accessible, non-judgmental, culturally, ethnically, and linguistically appropriate to the relevant populations, community-based, and independent of ability to pay or insurance/documentation status. They will also provide vital linkages to associated services, routine HIV testing, and primary health care.

In its initial pilot project, 2 community-based sites will serve as facilities at which patients may present for screening for post-exposure prophylaxis services, as well as sexually transmitted diseases. At the sites, initial eligibility and testing will be performed, and an initial 14-day supply of PEP medications will be provided if appropriate, and referrals will be initiated. All subjects who are provided an initial 14-day supply will be required to return to the site for the remainder of the 28-day course of medication, follow-up testing, adherence counseling, risk-reduction programming, and other appropriate referrals. Follow-up with patients by phone, email, and mobile-phone text message will be used as appropriate to maximize program retention.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age
* Able to understand and provide consent
* High-Risk Exposure Characteristic
* (one or more of the below, unprotected or with failed condom use)

  * Receptive Anal Intercourse
  * Insertive Anal Intercourse
  * Receptive Vaginal Intercourse
  * Insertive Vaginal Intercourse
* Receptive Oral Intercourse with Intraoral Ejaculation with known HIV+ source (supersedes all "high-risk source" criteria below)

  * Sharing injection drug works which have been intravascular
* High-Risk Source (one or more of the below)

  * Known HIV positive
  * MSM
  * MSM/W
  * IDU
  * CSW
  * Sexual perpetrator
  * From an endemic country (prevalence >1%)
  * Partner of one of the above
* Exposure within 72 hours of presentation
* Not known to be HIV positive
* No countermanding concomitant medications or allergies
* HIV-negative on presentation and without symptoms of PHI (do not withhold first dose pending these laboratory assessments).

Exclusion Criteria:

* Patients <18 years of age
* Unable to understand and provide consent
* Exposure >72 hours of presentation
* Known to be HIV positive
* Currently in-progress of a course of PEP initiated via non-P-QUAD mechanisms
* Any condition, which in the opinion of the intake provider, will seriously compromise the patient's ability to comply with the protocol, including

  * adherence to PEP medication dosing
  * Demonstrated HIV-positive on rapid testing
  * Unwillingness to commit to barrier-method (male and/or female condom) use until HIV-negative-status is confirmed 6 months after exposure
  * Unwillingness of breast-feeding women to transition to formula feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael J. Landovitz, M.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - L.A. Gay & Lesbian Center, Los Angeles, California
  - OASIS Clinic, Los Angeles, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two community-based sites, Jeffrey Goodman Clinic and The OASIS Clinic, will serve as facilities at which participants may present for screening for post-exposure prophylaxis services, as well as sexually transmitted diseases.
Groups:
- PEP Group: An intake of inclusion and exclusion criteria will be performed by program personnel. HIV-testing and STI testing will be provided as well as a brief and directed history and physical examination. If all inclusion and no exclusion criteria are met, an initial dose of PEP medications will be provided for immediate ingestion. A 14-day supply of PEP medications will be provided. Participant information sheets regarding PEP will be provided. Initial safety laboratory measurements and assessment of necessary referral services will be made, and behavioral risk assessment will stratify participants into "moderate behavioral risk," or "high behavioral risk." Moderate risk participants will receive risk-reduction programming within the P-QUAD program; high-risk participants will be referred externally to existing LA County behavioral risk-reduction programming.
Period: Overall Study
Arm/Group | PEP Group
Started | 267
Completed | 225
Not Completed | 42

BASELINE CHARACTERISTICS:
Arm/Group | PEP Group
Number analyzed (Participants) | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 266
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 32 [19 to 66]
Sex/Gender, Customized [Number; unit: participants]
  Male | 253
  Female | 11
  Transgender | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Black/AA | 23
  White | 128
  Hispanic/Latino(a) | 92
  Asian | 13
  American Indian/Alaska Native | 1
  Other | 10
Region of Enrollment [Number; unit: participants]
  United States | 267

OUTCOME MEASURES:

1. Primary Outcome: Retention, Measured as the Number of HIV Exposure Events That Were Retained in Care at the 24 Week Follow-up Visit
Time Frame: 24 Weeks
Population: 254 individuals were exposed to HIV once and received PEP; 11 individuals were exposed to HIV twice and received a PEP regimen twice; and 2 were exposed to HIV three times and received a PEP regimen for each of the three exposures
Measure: Count of Units; unit: HIV Exposure Events
Units Other Than Participants: HIV Exposure Events
Arm/Group | PEP Group
Number analyzed (Participants) | 267
Number analyzed (HIV Exposure Events) | 282
HIV Exposure Events
  Retained at 24 Weeks | 125
  Not Retained at 24 Weeks | 157
Statistical Analysis 1: Comparison: PEP Group; There was no power calculation for this analysis. The study was mainly descriptive, but Chi-square tests were used to determine if there were differences between individuals who were retained at the 24 Week Follow-up visit from individuals who were not retained at the 24 Week Follow-up visit; Test type: Other; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: Some individuals reenrolled in the study if an HIV exposure occurred at a later date. 254 individuals were exposed to HIV once and received PEP; 11 individuals were exposed to HIV twice and received a PEP regimen twice; and 2 were exposed to HIV three times and received a PEP regimen for each of the three exposures. A total of 282 PEP regimens were initiated on 267 unique individuals. 282 was used as the denominator for report Adverse Events.
Arm/Group | PEP Group
All-Cause Mortality (participants affected / at risk) | 0/282
Serious Adverse Events (participants affected / at risk) | 0/282
Other Adverse Events (participants affected / at risk) | 155/282
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEP Group (N=282)
Diarrhea (Gastrointestinal disorders) | 78
Nausea (Gastrointestinal disorders) | 48
Fatigue (General disorders) | 39
Mild to moderate abdominal discomfort (Gastrointestinal disorders) | 24

LIMITATIONS AND CAVEATS:
Open label clinical trial of deploying PEP regimens at community based sites. Non-randomized and guidelines have subsequently evolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No